CLINICAL TRIAL: NCT02128568
Title: A Feasibility Trial of the Youth Readiness Intervention: A Group Psychosocial Intervention for War-affected Youth in Sierra Leone
Brief Title: Sub-Trial of the Youth Readiness Intervention (YRI): Treatment of Control Group and Addition of Stress Biomarkers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Caritas Freetown (Other); McGill University (Other); Yale University (Other); The City College of New York (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Associate Professor of Child Health and Human Rights, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RPCGA-YRI-21003-Bio
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Anxiety Disorder; Depressive Disorder; Social Problems; Stress, Psychological; Violence, Non-accidental
Keywords: Depression/therapy;; Developing Countries;; Interpersonal Relations;; Life Change Events;; Psychotherapy, Group;; Resilience, Psychological;; Sierra Leone;; Survivors/psychology;; Social Adjustment;; Social Behavior;; War
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress, Psychological; Depression; Social Adjustment; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waitlist + YRI only (Active Comparator): Participants will complete the assessment and collection of biomarkers and be placed on a waitlist. Once the trial of the first arm has been concluded, participants complete another round of assessments and are offered the YRI sessions. The epigenetic biomarkers collected will be compared with the experimental arm.
  Interventions: Behavioral: Youth Readiness Intervention
- YRI only (Experimental): Immediately following assessment and collection of biomarkers, participants will be offered the YRI sessions.
  Interventions: Behavioral: Youth Readiness Intervention

INTERVENTIONS:
Behavioral: Youth Readiness Intervention — The YRI brings together six empirically-supported practice elements shown to be efficacious across different mental health interventions, as well as methods intended to socialize youth and improve self-efficacy. Practice elements address the broad scope of problems evidenced in Sierra Leonean war-affected youth and enhance the YRI's pacing, which progresses through three phases traditionally used in trauma treatments (stabilization, integration, connection). The weekly intervention takes place over 12 sessions lasting approximately one hour and a half. Groups are divided by gender and age. Each group is paired with two interventionists of the same gender.

SUMMARY:
This research is a continuation of the Youth Readiness Intervention (YRI) randomized clinical trial by adding additional pre and post intervention data collection upon treatment of the control group (N=222) with the intervention which was proven effective in the larger trial. The overall research has investigated whether participation in the YRI intervention will improve emotional regulation, prosocial attitudes/behavior, social support and daily and functioning among war-affected 15-24 year olds in Sierra Leone. In this sub-study which will involve treatment of the control group with the effective YRI intervention, the investigators will add an additional measure of self-regulation as observed via DNA methylation in buccal cells collected via cheek swabs. As before, after the YRI intervention, youth will be offered a free educational opportunity at the EducAid program in Freetown or in one of its upline/provincial sites. This stage of the research, as in the treatment with the main group, will test whether youth enrolled in the YRI psychosocial intervention go on to demonstrate improved attendance and behavior in a subsidized education program. In the previous phase of the trial, the investigators did observe significant effects for the YRI intervention and evidence that the program is indeed effective. For instance, post-intervention, YRI youth reported greater improvements in emotion regulation (β=0.109, 95%CI 0.026 to 0.191, δ=0.31), prosocial attitudes/behaviors (β=0.149, 95%CI 0.057 to 0.240, δ=0.38), and social support (β=0.119, 95%CI 0.009 to 0.229, δ=0.26) than controls, and greater reductions in functional impairments (β= -0.175, 95%CI -0.299 to -0.050, δ= -0.35). Differences in symptoms were non-significant at six-month follow-up for the full sample; moderator analyses showed that, for individuals in the top quartile of baseline symptoms, YRI youth had greater improvements in emotion regulation and social support than controls. At eight-month follow-up, teachers reported that YRI participants were 8.9 times more likely to be in school (28.8% v. 4.7%) and showed better attendance (β=3.553, 95%CI 0.989 to 6.118, OR=34.93) and academic performance (β= -0.954, 95%CI -1.807 to -0.102, δ= -1.31).

In this final phase of the trial as the investigators treat the wait list control group, the investigators will test whether intervention effects observed in self-report data on improved emotion-regulation are also upheld in biomarker data. Thus, the investigators will now provide YRI treatment to the wait list control group and employ the use of biomarkers as a measure of the intervention's effectiveness. The objective of the study will be to assess whether DNA methylation (collected via cheek swabs of buccal cells) is associated with changes in emotion regulation pre- and post- intervention. The aim is to test the hypothesis that the YRI is associated with improvements emotion-regulation evidence both in self-report data on emotion-regulation and in buccal cell DNA methylation. This study will add to the evidence base for effective, culturally sensitive mental health services for youth and young adults affected by war and other forms of adversity.

DETAILED DESCRIPTION:
In Sierra Leone, a dangerous gap remains between long-term psychosocial needs and adequate services. As youth affected by the war begin to enter adulthood, they face new challenges including unemployment, interrupted education, the need to support families, marginalization and stigma, as well as the remaining psychological effects of exposure to war. Healthy social integration is critical to the long-term wellbeing of this generation, but the evidence base on effective interventions to improve skills and self-efficacy is severely limited. Despite the high burden of mental health problems among war-affected youth in Sub-Saharan Africa, few empirically-supported behavioral treatments (ESBTs) or evidence-based interventions have been implemented in this region. This study stands to make an important contribution to knowledge on effective and culturally-sensitive mental health services that can be implemented in settings fraught by multiple hardships, including war, poverty, low educational attainment, and other hardships.

The Research Program on Children and Global Adversity at the Harvard School of Public Health has implemented the Youth Readiness Intervention (YRI) to address some of the challenges that youth face, including lack of education and employment, stigma and marginalization, and the long-term psychological effects of exposure to war. The YRI is an evidence-based group intervention designed to improve emotion regulation/reduce anger and foster prosocial functioning among 15-24 year old war-affected youth. It is grounded in findings from Betancourt et al.'s three wave-longitudinal study carried out from 2002 to 2008, which provides insight into how the adjustment of youth in post-conflict Sierra Leone is shaped by violence exposure and post -conflict loss and life disruption including family reconfiguration.

The intervention has three main goals: (1) Develop emotion regulation skills for healthy coping; (2) Develop problem solving skills to assist with achieving goals; (3) Improve interpersonal skills to enable healthy relationships and effective communication. Primary mental health outcomes include decreased anxiety, hostility, and depression, and increased pro-social attitudes, as measured by the Oxford Refugee Studies Psychosocial Adjustment Scale and the African Youth Psychosocial Assessment.

The addition of biomarkers research will build on a rare randomized controlled trial conducted in 2012-2014, where the control group will now receive the treatment and will be randomized in a lagged design to YRI or control and then all participants treated with the YRI. Therefore, the research data collection of the biomarkers will have three overarching aims: 1) To develop feasible and acceptable methods for collecting and analyzing genetic and epigenetic biomarkers from war-exposed youth in Sierra Leone. This will include forging collaborations with expert colleagues engaged in biomarker research, development of ethical protocols for data collection/storage, and review of the literature on genetic variation and mechanisms related to psychopathology. 2) To obtain biosamples from the control study participants of the randomized controlled YRI trial (2012-2014) and investigate the possibility of using this research methodology as a component of a fourth wave of data collection among war-affected youth and their families. 3) To investigate improvements in epigenetic marks (DNA methylation) pre- and post- the Youth Readiness Intervention and its associations with the findings from participants' self-reports on emotion regulation and prosocial functioning.

EducAid is a charitable trust established in 1994. Devoted to promoting education among underprivileged and war-affected young people in Sierra Leone through holistic and academic learning, EducAid provides free year-round education to over 1,500 youth, along with food, medicine, and shelter when needed. EducAid has a keen interest in exploring how psychosocial interventions can promote academic, social, and emotional well-being in students. EducAid's education model aims to improve academic knowledge, self-efficacy, and attitudes toward school. Additionally, it aims to nurture hope for the future and a sense of normalcy through interactions with teachers, mentors, and peers. Following participation in the education component, participants' employment and economic activity will be assessed using standardized instruments for cross-cultural work, including the World Bank Living Standards Surveys.

The Douglas Institute's Research Centre is the oldest centre of its kind in Quebec. With an annual budget of $18.5 million USD, it brings together over 300 distinguished researchers and post-doctoral fellows from all over the world, whose breakthroughs produce some 215 scientific publications every year. Recognized as a flagship centre by the Fonds de la recherche en santé du Québec (FRSQ), the provincial health research fund, the Research Centre, overseen by a board of directors, is financed in part by the Douglas Institute Foundation and in part by Canada's most prestigious research grants, including Canadian Institutes of Health Research (CIHR) and FRSQ, to name just two. It also sets itself apart with innovative research projects in the neurosciences, clinical and psychosocial divisions. In addition, the World Health Organization (WHO) Collaborating Centre in Montreal chose the Institute to establish its Centre for Research and Training in Mental Health.

ELIGIBILITY:
The control group of the YRI are the only eligible participants to complete the biomarkers .They were screened based on the eligibility requirements for the YRI, described below.

The screening tool contains four sections:

1. Consent and Age: assures that participants meet the age requirements
2. Oxford Refugees Psychosocial Adjustment Scale: assesses internalizing and externalizing problems in war affected youth and was developed and validated for use in Sierra Leone
3. Functioning: assesses the participant's ability to carry out activities of daily living
4. Psychological Analysis: clinician's assessment of the psychological state of the participant.

Inclusion Criteria:

* Participants must be from the control group of the YRI study; the inclusion criteria described below.

  * Participants must be between 15-24 years of age;
  * Participants must be school-intending at time of enrollment (2012)
  * A participant's total score on the Oxford scale must equal or exceed 30 AND
  * Participants must display at least one non-zero score on the functional impairment questions.

Exclusion Criteria:

* Participant does not plan to reside in the Freetown urban area for the duration of the study (9 months from start date);
* Participant fails to meet age requirements;
* Participant fails to meet Oxford psychosocial or functioning thresholds;
* Participant is judged by clinical staff as:

  o Needing mental health treatment beyond the scope of the YRI
* Otherwise not suitable for a cheek swab data collection.
* Participant displays the following:

  * Severe cognitive delays which preclude comprehension and ability to respond to items on the Youth Assessment Battery
  * Active suicidality
  * Psychosis
  * Risk of harm to themselves or others

Participants at risk of harm to themselves or others will be referred to local mental health or social work treatment facilities as appropriate.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Collection of epigenetic biomarker samples | Administered at 2 timepoints: (1) baseline; (2) within 15 days of YRI completion
  Description: Emotion regulation will be measured via epigenetic biomarkers, specifically DNA methylation of buccal cells collected via cheek swabs. A buccal cheek swab allows for rapid and consistent isolation of genomic DNA and is a convenient method for the acquiring of a DNA sample to examine methylation. DNA will be extracted for the purpose of identifying epigenetic marks (DNA methylation) across the genome and for sequence analysis of specific genomic regions. The DNA methylation data will be analyzed in relation to trauma history and intervention receipt, examining potential epigenetic changes associated with functionally relevant outcomes. Analysis of survey data will use inferential statistics to measure changes in constructs of relevance to the YRI, such as emotional regulation and perceived emotional, instrumental and informational support from others, community acceptance, and interpersonal skills.
Change in scores on the Oxford Measure of Psychosocial Adjustment & World Health Organization Disability Assessment Schedule, 2.0 (WHODAS 2.0) | Administered at 2 timepoints: (1) baseline; (2) within 15 days of YRI completion
  Primary outcomes of interest include the DERS (Disturbances in Emotion Regulation Scale), psychological distress (combined internalizing and externalizing problem scores) and changes in pro-social behaviors measured by the Oxford Refugee Studies Psychosocial Adjustment Scale. An additional primary outcome, daily functioning, will be assessed by the World Health Organization Disability Assessment Schedule, 2.0 (WHODAS 2.0). All measures are incorporated within the study's comprehensive Youth Assessment Battery.
Change in scores on the Youth Assessment Battery | Administered at 2 timepoints: (1) baseline; (2) within 15 days of YRI completion
  Secondary outcomes include the participant's interpersonal and community relations, experience of daily hardships, coping skills, post-traumatic stress, emotion regulation, health, risk behaviors, and other constructs as they relate to the YRI intervention areas.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, ScD, MA, Principal Investigator — Department of Global Health and Population, Harvard School of Public Health
Locations (1):
- CARITAS Freetown, Freetown, Sierra Leone

REFERENCES:
- [Background] Betancourt TS, Borisova II, de la Soudiere M, Williamson J. Sierra Leone's child soldiers: war exposures and mental health problems by gender. J Adolesc Health. 2011 Jul;49(1):21-8. doi: 10.1016/j.jadohealth.2010.09.021. Epub 2010 Dec 24. PMID 21700152
- [Background] Betancourt TS. Attending to the mental health of war-affected children: the need for longitudinal and developmental research perspectives. J Am Acad Child Adolesc Psychiatry. 2011 Apr;50(4):323-5. doi: 10.1016/j.jaac.2011.01.008. No abstract available. PMID 21421171
- [Background] Betancourt TS, Borisova II, Williams TP, Brennan RT, Whitfield TH, de la Soudiere M, Williamson J, Gilman SE. Sierra Leone's former child soldiers: a follow-up study of psychosocial adjustment and community reintegration. Child Dev. 2010 Jul-Aug;81(4):1077-95. doi: 10.1111/j.1467-8624.2010.01455.x. PMID 20636683
- [Background] Betancourt TS, Brennan RT, Rubin-Smith J, Fitzmaurice GM, Gilman SE. Sierra Leone's former child soldiers: a longitudinal study of risk, protective factors, and mental health. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):606-15. doi: 10.1016/j.jaac.2010.03.008. Epub 2010 May 1. PMID 20494270
- [Background] Betancourt TS, Agnew-Blais J, Gilman SE, Williams DR, Ellis BH. Past horrors, present struggles: the role of stigma in the association between war experiences and psychosocial adjustment among former child soldiers in Sierra Leone. Soc Sci Med. 2010 Jan;70(1):17-26. doi: 10.1016/j.socscimed.2009.09.038. Epub 2009 Oct 28. PMID 19875215
- [Background] Betancourt TS, Simmons S, Borisova I, Brewer SE, Iweala U, Soudiere MD. High Hopes, Grim Reality: Reintegration and the Education of Former Child Soldiers in Sierra Leone. Comp Educ Rev. 2008 Nov 1;52(4):565-587. doi: 10.1086/591298. No abstract available. PMID 19337570
- [Background] Betancourt TS, Bass J, Borisova I, Neugebauer R, Speelman L, Onyango G, Bolton P. Assessing local instrument reliability and validity: a field-based example from northern Uganda. Soc Psychiatry Psychiatr Epidemiol. 2009 Aug;44(8):685-92. doi: 10.1007/s00127-008-0475-1. Epub 2009 Jan 22. PMID 19165403
- [Background] Verdeli H, Clougherty K, Onyango G, Lewandowski E, Speelman L, Betancourt TS, Neugebauer R, Stein TR, Bolton P. Group Interpersonal Psychotherapy for depressed youth in IDP camps in Northern Uganda: adaptation and training. Child Adolesc Psychiatr Clin N Am. 2008 Jul;17(3):605-24, ix. doi: 10.1016/j.chc.2008.03.002. PMID 18558315
- [Background] Bolton P, Bass J, Betancourt T, Speelman L, Onyango G, Clougherty KF, Neugebauer R, Murray L, Verdeli H. Interventions for depression symptoms among adolescent survivors of war and displacement in northern Uganda: a randomized controlled trial. JAMA. 2007 Aug 1;298(5):519-27. doi: 10.1001/jama.298.5.519. PMID 17666672
- [Background] Betancourt TS, Speelman L, Onyango G, Bolton P. A qualitative study of mental health problems among children displaced by war in northern Uganda. Transcult Psychiatry. 2009 Jun;46(2):238-56. doi: 10.1177/1363461509105815. PMID 19541749
- [Background] Betancourt TS, Khan KT. The mental health of children affected by armed conflict: protective processes and pathways to resilience. Int Rev Psychiatry. 2008 Jun;20(3):317-28. doi: 10.1080/09540260802090363. PMID 18569183
- [Background] Betancourt TS. Child soldiers: reintegration, pathways to recovery, and reflections from the field. J Dev Behav Pediatr. 2008 Apr;29(2):138-41. doi: 10.1097/DBP.0b013e31816be946. No abstract available. PMID 18408537
- [Background] Betancourt TS, Williams T. Building an evidence base on mental health interventions for children affected by armed conflict. Intervention (Amstelveen). 2008;6(1):39-56. doi: 10.1097/WTF.0b013e3282f761ff. PMID 19997531